CLINICAL TRIAL: NCT06518473
Title: The Relation Between Atopy and Frequency of Exacerbation in Chronic Obstructive Pulmonary Disease Patients
Brief Title: Atopy and Frequency of Exacerbation in Chronic Obstructive Pulmonary Disease Patients
Status: Recruiting | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elmoniem Mohamed, Lecturer of chest medicine, Mansoura University Hospital
Other Study IDs: R.24.06.2680
Record Dates: First submitted 2024-07-14; First posted 2024-07-24 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: atopy; frequency of exacerbation; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Patch Tests

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic obstructive pulmonary disease patients: Adults aged 40-70 years diagnosed with COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2024 criteria
  Interventions: Diagnostic Test: Skin prick test

INTERVENTIONS:
Diagnostic Test: Skin prick test — Skin Prick Test (SPT): Common allergens including pollen, dust mites, Pet dander and mold.
  Serum IgE Levels: Total IgE Peripheral blood eosinophil was defined as an eosinophil count ≥ 5%, Quality of Life Assessment: COPD Assessment Test (CAT)
  Other Names: Total IgE

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a heterogeneous lung condition characterized by chronic respiratory symptoms (dyspnea, cough, sputum production and/or exacerbations) due to abnormalities of airways (bronchitis, bronchiolitis) and/or alveoli (emphysema) that cause persistent, often progressive, airflow obstruction.

The presence of non-fully reversible airflow obstruction (FEV1/FVC < 0.7 post-bronchodilation) measured by spirometry confirms the diagnosis of COPD

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease(COPD) is a heterogeneous lung condition characterized by chronic respiratory symptoms (dyspnea, cough, sputum production and/or exacerbations) due to abnormalities of airways (bronchitis, bronchiolitis) and/or alveoli (emphysema) that cause persistent, often progressive, airflow obstruction.

The presence of non-fully reversible airflow obstruction (FEV1/FVC < 0.7 post-bronchodilation) measured by spirometry confirms the diagnosis of COPD Inflammation of the bronchial wall is characterized by the presence of neutrophils and macrophages and by increased concentrations of IL-8 and Th1 cytokines, as well as by a proteinase /antiproteinase imbalance, and this could explain the poorer response to inhaled corticosteroids (ICs) seen in COPD.

Asthma may also be a risk factor for the development of chronic airflow obstruction and COPD and Epidemiological Study of Airway Obstructive Disease, adults diagnosed of asthma were found to have a 12-fold higher risk of acquiring COPD over time compared to those without asthma, after adjusting for smoking.

Although both COPD and asthma are associated with chronic inflammation of the respiratory tract, there are differences in the inflammatory cells and mediators involved in the two diseases, some patients with COPD have an inflammatory pattern with increased eosinophils cells, similar to that of asthma.

When there is diagnostic of Asthma and COPD overlap (ACO) uncertainty, an elevated total serum immunoglobulin E (IgE; >100 international units/mL), elevated peripheral blood eosinophil count (>300 cells/microL), and evidence of allergic disease (eg, skin testing or immunoassays for perennial allergen sensitivity) may point a clinician to asthma or Asthma - COPD overlap (ACO). Elevated sputum eosinophil counts, if available, are more common in asthma or ACO than COPD The Dutch hypothesis suggests that atopy and bronchial hyper-responsiveness , which are important markers of asthma, can be involved in the pathogenesis of COPD, although there is no clear evidence regarding the frequency of atopy (including asthma), Allergic rhinitis (AR), eczema, or increased IgE levels in patients with COPD, because most studies have involved small samples and limited evaluation of atopy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-70 years diagnosed with COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2024 criteria

Exclusion Criteria:

* Patients with known allergic diseases before enrollment
* Patients with associated other chronic respiratory disorders
* Patients with significant comorbidities that could influence respiratory function.
* Recent respiratory infections or use of systemic corticosteroids within the last month before enrollment.

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults aged 40-70 years diagnosed with COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2024 criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-14 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Atopy in chronic obstructive pulmonary disease patients | 6 months
  Total IgE (mg/dl) and ) will be assessed in chronic obstructive pulmonary disease patients
Chronic obstructive pulmonary disease patients | 2 months
  Blood eosinophil count (%) will be assessed in chronic obstructive pulmonary disease patients

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, lecturer, Principal Investigator — Lecturer of chest medicine Faculty of medicine Mansoura university
Locations (1):
- Mohamed AbdElmoniem, Al Mansurah, Egypt